CLINICAL TRIAL: NCT07175402
Title: Development, Feasibility, Efficacy, and Cost-effectiveness of an Online ACT Intervention for Disorders of Gut-Brain Interaction (Beta Trial)
Brief Title: Feasibility and Acceptability of an Online ACT Intervention for Disorders of Gut-Brain Interaction - Beta Trial
Acronym: iACTforDGBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: Sahlgrenska University Hospital (Other); Göteborg University (Other); Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-00751d
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: DGBI; Depression/Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: This is a second (beta) pilot study (feasibility including acceptability) in which the investigators intend to see how the intervention and overall workload (including measurements) is perceived by the participants.
Who Masked: Participant
Masking Description: Principal Investigator, other investigators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy (ACT) (Experimental): Acceptance and Commitment Therapy (ACT)
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)
- Education on DGBI, psychoeducation (Active Comparator): Education on DGBI, psychoeducation
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — The Online version of Acceptance and Commitment Therapy (iACTforDGBI) intervention will include 8 weekly sessions of around 20 minutes each, and will comprise ACT-consistent informative texts, audio exercises, and videos. The intervention is expected to have the following overall structure: Session 0: Individual videoconference meeting, introduction. Session 1: Creative hopelessness and mindfulness. Session 2: The body, acceptance, and values. Session 3: Compassion. Session 4: Cognitive defusion and committed action. Session 5-7: Personalised content (in-depth material and tasks based on individual difficulties assessed with diary). Session 8: Summary of intervention.
  Arms: Acceptance and Commitment Therapy (ACT)
Other: Psychoeducation — Participants in the active control group will be asked to complete 8 weekly 20-minute sessions of an online course for education on DGBIs. This course will be delivered through a similar platform than the one delivering the online ACT for DGBI intervention, via the same website. The intervention platform will have similar designs and structure, and will be developed by the same web development company. Session 0: Individual session, introduction. Session 1-8: The content will be based on the IBS school intervention (e.g., Ringström et al., 2009), in particular its online version (Lindfors et al., 2021), developed by members of the current research team. This education intervention was based on the biopsychosocial model of DGBI and was originally developed and tested as a face-to-face group intervention with six 2-h sessions held weekly. IBS school generally aims at increasing disease knowledge in people with IBS and covers a wide spectrum of issues related to IBS.
  Arms: Education on DGBI, psychoeducation

SUMMARY:
The goal of this clinical trial is to assess the acceptability, feasibility, and usability of the iACTforDGBI intervention among patients with Disorders of Gut-Brain Interaction (DGBI). The main question it aims to answer are:

What are the perceptions of patients with DGBI and healthcare practitioners regarding the acceptability, feasibility, and usability of the iACTforDGBI intervention?

Participants will be asked to:

Complete the iACTforDGBI intervention prototype, consisting of self-guided online sessions.

Participate in online interviews and fill out online questionnaires to evaluate the intervention concerning acceptability, feasibility, usability and preliminary effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years
2. Meeting clinical symptom levels for least one DGBI diagnosis (assessed with the Rome IV Diagnostic Questionnaire for Functional Gastrointestinal Disorders in Adults (Palsson et al., 2016))
3. Clinically meaningful levels of depressive symptoms or anxiety: score ≥ 13 on the Montgomery Åsberg Depression Rating Scale (MADRS-S; depressive symptoms), or score ≥ 10 on the Generalized Anxiety Disorder scale-7 (GAD-7; anxiety symptoms; Spitzer et al., 2006)
4. Stable medication for psychiatric symptoms including anxiety, depression and sleep problems for at least two months prior to intervention.
5. Ability to read and write Swedish
6. Have access to a device (like computer, tablet or smartphone with) with access to the internet and that can be used to attend video conferences and preview the intervention platform (i.e., have a microphone and speakers or headphones).

Exclusion Criteria:

1. Currently undergoing any form of psychological intervention.
2. Increased risk of suicide (≥4 points on MADRS item 9)
3. Severe depression (≥34 points on MADRS)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Individual interviews | At post treatment (8 weeks)
  Feasibility and acceptability of intervention

SECONDARY OUTCOMES:
The Generalized Anxiety Disorder scale-7 (GAD-7) | At pre and post treatment (0 and 8 weeks).
  Symptoms of general anxiety, min-max: 0-21, higher scores: more symptoms of general anxiety.
EQ-5D-5L | At pre and post treatment (0 and 8 weeks)
  Health-related Quality of Life, min-max 0-1 (index value), higher scores: better health-related quality of life
AQoL-8D | At pre and post treatment (0 and 8 weeks)
  Health-related Quality of Life, min-max -0.04-1.00, higher scores: better health-related quality of life.
The Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry (TIC-P) | At pre and post treatment (0 and 8 weeks)
  Healthcare Utilization, no fixed range (reports number of contacts, costs etc.), higher scores: greater healthcare utilization/higher costs.
The Gastrointestinal Symptom Rating Scale (GSRS) | At pre and post treatment (0 and 8 weeks)
  Symptom Severity of DGBI, min-max 19-133, higher scores: more severe gastrointestinal symptoms.
The Chronic Illness Shame Scale (CISS) | At pre and post treatment (0 and 8 weeks)
  Shame of Chronic Illnesses, min-max 0-28, higher scores: greater shame related to chronic illness.
The Credibility/Expectancy Questionnaire (CEQ) | After session 2 (2 weeks)
  Treatment Credibility and Expectancy, min-max 0-27 credibility, 0-9 expectancy, higher scores: higher treatment credibility/expectancy.
The System Usability Scale (SUS), min-max 0-100, higher scores: greater perceived usability. | At post treatment (8 weeks)
  Intervention Platform Usability
The Negative Effects Questionnaire (NEQ-20), min-max 0-80 (depending on number of endorsed negative effects), higher scores: more negative effects/adverse events. | At post treatment (8 weeks)
  Negative side effects and events
The Intervention Acceptability Scale | At post treatment (8 weeks)
  Intervention Acceptability, min-max 1-5 per item, higher scores: greater intervention acceptability.
The Contextual Therapies Process Awareness Scale | At post treatment (8 weeks)
  Awareness of Processes, min-max 1-5 per item, higher scores: greater process awareness.
The Patient Health Questionnaire-9 (PHQ-9) | At pre and post treatment (0 and 8 weeks)
  Symptoms of depression, min-max 0-27, higher scores: more depressive symptoms.
The Multidimensional Psychological Flexibility Inventory (MPFI) | At pre and post treatment (0 and 8 weeks)
  Psychological flexibility, min-max 1-6 per item, higher scores: indicate more rigidity/avoidance on negative sub scales
The State Self-Compassion Scale - short form (SSCS-S) | At pre and post treatment (0 and 8 weeks)
  State self-compassion, min-max 6-30, higher scores: greater state self-compassion.
The Self-Compassion Scale - short form (SCS-SF) | At pre and post treatment (0 and 8 weeks)
  Trait self-compassion, min-max 12-60, higher scores: greater trait self-compassion.

CONTACTS AND LOCATIONS:
Locations (1):
- Örebro University, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
This question is under investigation. Some of the data contain sensitive information on health, and the main priority is participants integrity which need to be balanced against basic scientific principles on scrutiny. However, any personal data that can be shared without compromising participants integrity to a reasonable degree will be shared upon reasonable request.